CLINICAL TRIAL: NCT02894554
Title: A Single-Center, Open-Label Study to Evaluate the Renal Function Improvement in Lamivudine Long Term Used HBsAg Positive Kidney Transplantation Patients After Switch to Telbivudine Treatment.
Brief Title: Renal Function Improvement in HBsAg Positive Kidney Transplantation Patients Under Telbivudine Treatment.
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: clinical myalgia
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 201310070MINA
Record Dates: First submitted 2015-07-07; First posted 2016-09-09 (Estimated); Last update posted 2016-09-09 (Estimated); Status verified 2016-09

CONDITIONS: HBsAg-positive Renal Allograft Recipients
MeSH Terms: interventions — Telbivudine; Lamivudine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- lamivudine (Placebo Comparator): HBsAg (+) patients received renal transplant and under lamivudine therapy.
  Interventions: Drug: Lamivudine
- telbivudine (Active Comparator): HBsAg (+) patients received renal transplant and under lamivudine therapy and then switch to telbivudine 6 months later.
  Interventions: Drug: Telbivudine

INTERVENTIONS:
Drug: Telbivudine
  Other Names: Sebivo
  Arms: telbivudine
Drug: Lamivudine
  Other Names: Zeffix
  Arms: lamivudine

SUMMARY:
The hepatitis B virus (HBV) infection rate among renal transplant recipients was reported from 3% to 20.9%. And patient survival and graft survival rates following renal transplantation may be worsen in HBsAg-positive carriers than in HBsAg-negative recipients. Due to viral replication in asymptomatic HBV carriers induced by post-transplant immunosuppression, liver-related complications, such as liver failure and bleeding, account for 37% to 57% of the mortality cases in HBsAg-positive renal allograft recipients.

Since the late 1990s, Lamivudine has been recognized as an effective and well-tolerated antiviral drug for chronic HBV infection. Lamivudine treatment among HBsAg-positive renal allograft recipients has significantly improved patient survival rates during short-term follow-up. Telbivudine is another approved nucleoside antiviral agent for patients with chronic hepatitis B (CHB). Recently, it was shown that eGFR was improved in HBV-related decompensated cirrhosis patients after 52 weeks Telbivudine treatments. Additional eGFR increase was also observed in Lamivudine experienced CHB patients after switch to Telbivudine treatment.

However, limited results were known about the renal function affected by oral anti-HBV drugs when patients received kidney transplantation. Therefore, we would like to conduct this study to evaluate the renal function of Lamivudine long term used HBsAg positive patients received kidney transplantation after switch to Telbivudine treatment. The clinical and virological outcomes will provide valuable insights of clinical practice.

ELIGIBILITY:
Inclusion Criteria:

1. Kidney transplant patients who are treated with Lamivudine over 6 months (Considering include post kidney transplantation > 6 months with stable calcineurin inhibitors level
2. Seropositive of HBsAg for 6 months
3. Willing and able to provide written informed consent

Exclusion Criteria:

1. Hepatitis cirrhosis patients
2. Co-infection with hepatitis C virus or HIV
3. Pregnant or nursing
4. YMDD resistant at baseline
5. ABO incompatible renal transplantation
6. Cross match positive
7. Poor renal function at baseline (eGFR<20)
8. Known hypersensitivity or intolerance to any of the ingredients in Telbivudine
9. Known history of Telbivudine resistance

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2014-07; Primary Completion 2014-10 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
To evaluate the renal function in HBsAg positive kidney transplant patients in Telbivudine and Lamivudine treatment groups by eGFR at 48 Weeks after treatment using MDRD formula. | 48 weeks

IPD SHARING:
Plan to Share IPD: Yes